CLINICAL TRIAL: NCT01992380
Title: Test-Retest Reproducibility of 18F-AV-1451 Injection for Brain Imaging of Tau in Healthy Volunteers and Cognitively Impaired Subjects.
Brief Title: A Study of Flortaucipir PET in Healthy Volunteers and Cognitively Impaired Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A03
Record Dates: First submitted 2013-11-08; First posted 2013-11-25 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy Volunteer Subjects (Experimental): Healthy males or females 50 years or older with no evidence of cognitive impairment
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET scan
- MCI subjects (Experimental): Subjects 50 years or older with mild cognitive impairment (MCI)
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET scan
- Probable AD Subjects (Experimental): Subjects 50 years or older with probable Alzheimer's Disease (AD)
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET scan

INTERVENTIONS:
Drug: Flortaucipir F18 — IV injection, 370 MBq (10 mCi), two doses up to four weeks apart
  Other Names: [F18]T807; 18F-AV-1451; Tauvid
Procedure: Brain PET scan — positron emission tomography (PET) scan of the brain at 80-100 and 110-130 minutes after injection

SUMMARY:
This study will test if two flortaucipir PET scans up to 4 weeks apart in healthy volunteers, MCI and AD subjects provide the same results.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers

  * Male or female subjects ≥ 50 years of age
  * Mini-mental state examination (MMSE) ≥ 29
* MCI Subjects

  * Male or female subjects ≥ 50 years of age
  * MMSE ≥ 24
  * Have MCI consistent with National Institute on Aging-Alzheimer's Association (NIA-AA) working group's diagnostic guidelines for AD
  * Have a study partner that can report on subject's activities of daily living
* Probable AD Subjects

  * Male or female subjects ≥ 50 years of age
  * MMSE > 10
  * Meet clinical criteria for probable AD based on the NIA-AA working group's diagnostic guidelines for AD
  * Have a study partner that can report on subject's activities of daily living

Exclusion Criteria:

* Current clinically significant psychiatric disease
* Evidence of structural brain abnormalities
* Evidence of dementing illness other than AD
* Current clinically significant cardiovascular disease or ECG abnormalities, or additional risk factors for Torsades de Pointes
* Current clinically significant infectious disease, endocrine or metabolic disease, pulmonary, renal or hepatic impairment, or cancer
* History of alcohol or substance abuse or dependence
* Females of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception
* Have received or participated in a trial with investigational medications in the past 30 days
* have had a non-study related radiopharmaceutical imaging or treatment procedure within 7 days prior to the study imaging session.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-11-13 (Actual); Primary Completion 2014-05-30 (Actual); Study Completion 2014-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Chair — Avid Radiopharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Research Site, Newport Beach, California
  - Research Site, New Haven, Connecticut

REFERENCES:
- [Result] Devous MD Sr, Joshi AD, Navitsky M, Southekal S, Pontecorvo MJ, Shen H, Lu M, Shankle WR, Seibyl JP, Marek K, Mintun MA. Test-Retest Reproducibility for the Tau PET Imaging Agent Flortaucipir F 18. J Nucl Med. 2018 Jun;59(6):937-943. doi: 10.2967/jnumed.117.200691. Epub 2017 Dec 28. PMID 29284675

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment between Nov 2013 and May 2014
Groups:
- Healthy Volunteer Subjects: Healthy males or females 50 years or older with no evidence of cognitive impairment
  Flortaucipir F18: IV injection, 370 MBq (10 mCi), two doses up to four weeks apart
  Brain PET scan: positron emission tomography (PET) scan of the brain
- MCI Subjects: Subjects 50 years or older with mild cognitive impairment (MCI)
  Flortaucipir F18: IV injection, 370 MBq (10 mCi), two doses up to four weeks apart
  Brain PET scan: positron emission tomography (PET) scan of the brain
- Probable AD Subjects: Subjects 50 years or older with probable Alzheimer's Disease (AD)
  Flortaucipir F18: IV injection, 370 MBq (10 mCi), two doses up to four weeks apart
  Brain PET scan: positron emission tomography (PET) scan of the brain
Period: Overall Study
Arm/Group | Healthy Volunteer Subjects | MCI Subjects | Probable AD Subjects
Started | 6 | 8 | 10
Completed | 6 | 8 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteer Subjects | MCI Subjects | Probable AD Subjects | Total
Number analyzed (Participants) | 6 | 8 | 10 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (9.5) | 70.3 (5.4) | 74.4 (7.3) | 70.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 2 | 8
  Male | 2 | 6 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 8 | 10 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 5 | 8 | 10 | 23
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 8 | 10 | 24
Mini Mental Status Exam (MMSE) [Mean (Standard Deviation); unit: units on a scale] — Mini-mental status exam (MMSE) is a 30-point questionnaire that is used to measure cognitive impairment. Scores range from 0 to 30 with lower scores representing greater levels of cognitive impairment.
  units on a scale | 29.7 (0.52) | 28.3 (1.58) | 23.9 (4.58) | 26.8 (3.95)

OUTCOME MEASURES:

1. Primary Outcome: Test-Retest Reproducibility
Description: Evaluate test-retest reproducibility of flortaucipir for brain imaging of tau in healthy volunteers and subjects with cognitive impairment. Standard uptake value ratios (SUVRs) for each scan, normalized to the cerebellar crus. A combination volume of interest (VOI) = weighted average of parietal, temporal, and occipital regions was used. The protocol pre-specified that test-retest endpoint was to be calculated for the combined group of healthy volunteers and cognitively impaired subjects
Time Frame: 80-100 minutes postdose
Population: All subjects with a valid test and re-test scan. The 80-100 minute scan was not done for one subject in the healthy volunteer group due to technical difficulties with the scanning apparatus
Measure: Mean (Standard Deviation); unit: standardized uptake value ratio (SUVr)
Groups:
- All Subjects: All study subjects
  Flortaucipir F18: IV injection, 370 MBq (10 mCi), two doses up to four weeks apart
  Brain PET scan: positron emission tomography (PET) scan of the brain
Arm/Group | All Subjects
Number analyzed (Participants) | 24
standardized uptake value ratio (SUVr)
  Test Imaging | 1.342 (0.341)
  Retest Imaging: number analyzed (Participants) | 23
  Retest Imaging | 1.355 (0.309)
Statistical Analysis 1: Comparison: All Subjects; Intraclass correlation coefficient [ICC(2,1)] analysis from Shrout and Fleiss; Test type: Other; ICC = 0.971, 95% CI 2-sided [0.935 to 0.988] — Assessed the agreement between the test and retest imaging of the combination VOI SUVr

2. Primary Outcome: Test-Retest Reproducibility
Description: Evaluate test-retest reproducibility of 18F-AV-1451 for brain imaging of tau in healthy volunteers and subjects with cognitive impairment. Standard uptake value ratios (SUVRs) for each scan, normalized to the cerebellar crus. A combination volume of interest (VOI) = weighted average of parietal, temporal, and occipital regions was used. The protocol pre-specified that test-retest endpoint was to be calculated for the combined group of healthy volunteers and cognitively impaired subjects
Time Frame: 110-130 minutes postdose
Measure: Mean (Standard Deviation); unit: standardized uptake value ratio (SUVr)
Arm/Group | All Subjects
Number analyzed (Participants) | 24
standardized uptake value ratio (SUVr)
  Test Imaging | 1.459 (0.455)
  Retest Imaging | 1.457 (0.396)
Statistical Analysis 1: Comparison: All Subjects; Intraclass correlation coefficient [ICC(2,1)] analysis from Shrout and Fleiss; Test type: Other; ICC = 0.968, 95% CI 2-sided [0.926 to 0.986] — Assessed the agreement between the test and retest imaging of the combination VOI SUVr

ADVERSE EVENTS:
Time Frame: End of study for AE reporting was 48 hours after flortaucipir administration at each imaging visit.
Description: Adverse Events were defined as occurring or worsening after injection of dose, within 48 hours post injection, at an imaging visit. AEs occurring after study drug administration, but outside that window were not recorded, unless considered attributable to flortaucipir.
Arm/Group | Healthy Volunteer Subjects | MCI Subjects | Probable AD Subjects
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 1/6 | 0/8 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteer Subjects (N=6) | MCI Subjects (N=8) | Probable AD Subjects (N=10)
dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less